CLINICAL TRIAL: NCT06770569
Title: Safety, Tolerability, and Pharmacokinetics of HRS-3802 Monotherapy in Patients With Malignant Solid Tumors: a Single-arm, Open, Multicenter Phase I Study
Brief Title: Safety, Tolerability, and Pharmacokinetics of HRS-3802 Monotherapy in Patients With Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-3802-101
Record Dates: First submitted 2024-12-26; First posted 2025-01-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-3802 (Experimental)
  Interventions: Drug: HRS-3802

INTERVENTIONS:
Drug: HRS-3802 — HRS-3802

SUMMARY:
The study is being conducted to evaluate the safety and tolerability of HRS-3802 monotherapy in patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be willing to participate in the study, sign the informed consent form, have good compliance, and cooperate with follow-up visits;
2. Age ≥18 years, male or female;
3. Patients with advanced malignant tumors confirmed pathologically;
4. Failure of adequate standard treatment, or no effective standard treatment;
5. Patients must have at least 1 extracranial measurable target lesion per RECIST v1.1;
6. The expected survival period is more than 12 weeks;
7. The Eastern Cooperative Oncology Group (ECOG) physical fitness score is 0 - 1;
8. Have sufficient bone marrow and organ function (have not received blood transfusion or hematopoietic stimulating factor treatment within 14 days);
9. Female subjects of childbearing age must undergo a serum pregnancy test within 7 days before starting the study medication, and the result is negative, and are willing to use a medically approved high-efficiency contraception during the study period and within 1 months after the last administration of the study drug Measures.

Exclusion Criteria:

1. Subjects had cancerous meningitis or untreated central nervous system metastases;
2. Subjects had severe cardiovascular and cerebrovascular diseases;
3. There is third-space effusion that cannot be controlled by drainage and other methods (such as massive ascites, pleural effusion, pericardial effusion);
4. Subjects had or currently had idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia , drug pneumonia, or CT during screening showed active pneumonia;
5. Arteriovenous thrombosis occurred within 6 months prior to the first dose;
6. Severe infection occurred within 4 weeks prior to initial administration;
7. Subjects with refractory nausea, vomiting, or other gastrointestinal disorders that affect the use of oral medications: including malabsorption syndrome;
8. Known history of human immunodeficiency virus (HIV) seropositive status or acquired immunodeficiency syndrome (AIDS);
9. Subjects had active hepatitis;
10. Subjects were scheduled to receive other systemic antitumor therapies during the study period;
11. Known allergies and contraindications to the investigational drug or any of its components;
12. Other factors as judged by the investigator that may lead to the termination of the study, such as other serious diseases, serious laboratory test abnormalities, or family or social factors that could affect the safety of the subject, or the collection of study data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events and the severity of adverse events | Every 4 weeks after treatment initiation (through study completion，an average 5 mouths)
Dose-limiting toxicity (DLT) | During the first 28-day cycle of HRS-3802 treatment
Maximum tolerated dose (MTD) | 3 weeks after treatment initiation
Recommended Phase II Dose (RP2D) | 3 weeks after treatment initiation

SECONDARY OUTCOMES:
Objective response rate (ORR) - RECIST 1.1 | Up to approximately 6 months
  ORR is defined as the proportion of subjects who have achieved complete response (CR) or partial response (PR) according to RECIST 1.1.
Duration of Response (DoR) per RECIST 1.1 | Up to approximately 2 years
Progression-free survival (PFS) per RECIST 1.1 | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (5):
  - GenesisCare North Shore (Oncology), Saint Leonards, New South Wales
  - Macquarie University Hospital, Sydney, New South Wales
  - John Flynn Private Hospital, Tugun, Queensland
  - GenesisCare St Andrews, Adelaide, South Australia
  - Peninsula and South Eastern Haematology & Oncology Group, Frankston, Victoria
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided